CLINICAL TRIAL: NCT01242085
Title: Alignment of Total Knee Components Using Standard or Custom Instrumentation
Brief Title: Preoperative Alignment of Total Knee Replacement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Principal Investigator, steven woolson, staff surgeon, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04061991
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Results first posted 2013-05-08 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Knee Arthritis
Keywords: alignment
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Active Comparator): control group will have standard instrumentation of their knee replacement
  Interventions: Procedure: control group
- trumatch group (Experimental): the trumatch patient will have custom instruments made from preop CT scans
  Interventions: Procedure: trumatch group

INTERVENTIONS:
Procedure: trumatch group — these patient will have CT based customized knee instruments used for surgery
  Other Names: trumatch CPI
  Arms: trumatch group
Procedure: control group — these patients will have standard instrumentation used for for knee replacement
  Other Names: Depuy knee instruments
  Arms: control group

SUMMARY:
The hypothesis of this study is that total knee alignment will be improved by preoperative planning from CT scans and the production of custom instruments compared to the use of standard instruments.

DETAILED DESCRIPTION:
Patients will be randomized to have either customized knee instruments or standard generic instrumentation for primary total knee replacement. Postoperative CT scan will be used to determine alignment of each group.

ELIGIBILITY:
Inclusion Criteria:patients undergoing primary total knee replacement -

Exclusion Criteria:patients who have hardware involving the hip, knee or ankle

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-11; Primary Completion 2012-05 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Palo Alto VA HCS, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 6-2010 thru 6-2011 at the VA Palo Alto HCS
Pre-assignment Details: 1 participant was excluded because withdrew prior to assignment
Groups:
- Trumatch Group: trumatch group will have customized knee instruments : CT based customized knee instruments
- Both Interventions: one participant had both interventions - one for each knee
Period: Overall Study
Arm/Group | Trumatch Group | Control Group | Both Interventions
Started | 30 | 33 | 1
Completed | 22 (8 patients did not undergo intervention since 4 had medical problems and 4 withdrew) | 26 (7 patients did not receive allocated intervention since 5 had medical problems and 2 withdrew) | 1
Not Completed | 8 | 7 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 0
Not completed — medically unable to have surgery | 4 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: control group will have standard instrumentation of their knee replacement: standard instrumentation for knee replacement
  study group will have customized knee instruments : CT based customized knee instruments
- Trumatch Group: patients randomized to study instrumentation
- Both Interventions: one participant had bilateral knee replacement with one control knee and one trumatch knee
- Total: Total of all reporting groups
Arm/Group | Control | Trumatch Group | Both Interventions | Total
Number analyzed (Participants) | 33 | 30 | 1 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 0 | 39
  >=65 years | 13 | 11 | 1 | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 65.1 (8.3) | 67.3 (7.7) | 81 (0) | 66.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 33 | 30 | 1 | 64
Region of Enrollment [Number; unit: participants]
  United States | 33 | 30 | 1 | 64
knee replacement participant [Number; unit: participants] | 33 | 30 | 1 | 64

OUTCOME MEASURES:

1. Secondary Outcome: Surgical Time
Description: the difference between the average surgical time will be determined and compared with 95% CI
Time Frame: intraoperative surgical time
Population: particpants who completed study
Measure: Mean (95% Confidence Interval); unit: delta between means in minutes
Arm/Group | Control | Trumatch Group
Number analyzed (Participants) | 26 | 22
delta between means in minutes | 4.0 [-2.1 to 10.2] | 0 [-2.1 to 10.2]

2. Primary Outcome: Alignment of Knee - Measured Mechanical Axis From CT Data
Description: the mean knee mechanical axis was determined from 3D CT data - negative value designates varus alignment
Time Frame: postoperatively - CT done within 1 week of surgery
Population: all participants who completed the study
Measure: Mean (95% Confidence Interval); unit: degrees
Arm/Group | Control | Trumatch Group
Number analyzed (Participants) | 26 | 22
degrees | -1.7 [-3.0 to -0.4] | -1.3 [-2.5 to -0.2]

ADVERSE EVENTS:
Arm/Group | Control | Trumatch Group
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/22
Other Adverse Events (participants affected / at risk) | 0/26 | 0/22

LIMITATIONS AND CAVEATS:
none except small sample sizes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No